CLINICAL TRIAL: NCT02349373
Title: The Focus of a Running Schedule and Its Association With the Risk of Running Injuries? A Randomized Trial.
Brief Title: Focus of a Running Schedule and Risk of Running Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-20140069
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Running Related Injuries
Keywords: Overuse injury; Running related injury; Running pattern
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preconditioning running (Active Comparator): An 8 week preconditioning period. The variables of interest are running distance and running intensity: running speed >80% VO2max (maximal oxygen uptake).
  Interventions: Behavioral: An 8 week preconditioning period
- Follow-up period (Active Comparator): The Volume group progress 23% in total weekly running distance in the last adaptation week in the prior 4 week block.
  The Intensity group progress 23% in weekly distance of running above 80% VO2 max (maximal oxygen uptake), based on the distance of running above 80% VO2max in the last adaptation week in the prior 4 week block.
  Interventions: Behavioral: 16 week training period

INTERVENTIONS:
Behavioral: An 8 week preconditioning period — Receipt of a weekly running schedule through an online training diary.
  Arms: Preconditioning running
Behavioral: 16 week training period — Receipt of a weekly running schedule through an online training diary.
  Arms: Follow-up period

SUMMARY:
Running is a natural part of human locomotion and humans have been running for million of years. In modern society, running has become a popular way of exercise and is undertaken by many people worldwide, possibly because it provides a cheap and easily accessible form of exercise, and the positive effects of running on health and fitness are well known. Unfortunately, running is also associated with a high risk of injury.

The purpose of this project is to investigate how a running schedule which focuses either on running distance or running speed influence the overall risk of injury and the types of injury sustained in recreational runners.

DETAILED DESCRIPTION:
Trails directed at investigating differences in injury risk in relation to the focus of the running schedule have been conducted without any firm conclusions. People engaged in recreational running or choosing running as a new and active lifestyle needs guidance on which running schedules minimize the injury risk, aiding their chance of an active lifestyle and possibly reversing the increase in people developing a lifestyle disease. To develop running schedules minimizing the risk of injury, an understanding of the mechanisms that the different training variables impose on the human body is necessary. The existing literature on running intensity and the development of injuries show conflicting result. More studies are necessary to ascertain if there is a relationship between the intensity of running. In such studies, it is important to include other training variables in the analysis and to quantify running exposure using an objective method of measuring the relative intensity and absolute volume.

ELIGIBILITY:
Inclusion Criteria:

* on average 1-3 weekly running sessions the past 6 months
* owns a pair of running shoes
* internet access and mail address
* owns a Garmin GPS watch (pulse rate watch) or an IPhone/Android phone

Exclusion Criteria:

* previous injury in lower extremity within the past 6 months
* unable to follow the running regime in 6 consecutive months
* do not want to use GPS (Global Positioning System) watch or Android/Smart phone to register training
* unable to read or understand Danish
* deprecated by personal GP (General Practitioner) to run due to former surgery or physical disease
* mental condition that does not allow participation (e.g. externalizing behaviors, dementia)
* pregnancy
* participants with blood pressure above normal according to WHO guidelines will need to consult own GP (General Practitioner) for approval

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Running Related Injury (RRI) | 24 weeks
  An injury will be reported through the online training diary. If the runners are injured an appointment for clinical examination is made with the diagnostic staff.

SECONDARY OUTCOMES:
Symptoms of overuse injury | 24 weeks
  A physical problem perceived as pain, tenderness, stiffness, aching, looseness and instability in any part of the body.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, M.D., Study Chair — Aalborg University Hospital; Daniel R. Joergensen, PhD student, Principal Investigator — University of Aarhus
Locations (1):
- Clinic for Neuro- and Orthopaedic Diseases, Aalborg University Hospital, Aalborg, Denmark

REFERENCES:
- [Derived] Ramskov D, Nielsen RO, Sorensen H, Parner E, Lind M, Rasmussen S. The design of the run Clever randomized trial: running volume, -intensity and running-related injuries. BMC Musculoskelet Disord. 2016 Apr 23;17:177. doi: 10.1186/s12891-016-1020-0. PMID 27107810